CLINICAL TRIAL: NCT02145260
Title: Randomized Trial of Dialysate Sodium in Chronic Hospitalized Hemodialysis Patients
Brief Title: Trial of Dialysate Sodium in Chronic Hospitalized Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Finnian McCausland, Assistant Professor of Medicine, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014P000629
Record Dates: First submitted 2014-05-13; First posted 2014-05-22 (Estimated); Results first posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Intra-dialytic Hypotension
Keywords: Hemodialysis; Hypotension; Hospitalization
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lower dialysate sodium (Active Comparator): Dialysate sodium concentration of 138 mmol/L
  Interventions: Drug: Lower dialysate sodium (138 mmol/L; using Renasol hemodialysis concentrate)
- Higher dialysate sodium (Experimental): Dialysate sodium concentration of 142 mmol/L
  Interventions: Drug: Higher dialysate sodium (142 mmol/L; using Renasol hemodialysis concentrate)

INTERVENTIONS:
Drug: Lower dialysate sodium (138 mmol/L; using Renasol hemodialysis concentrate) — A lower dialysate sodium will bes used in the active comparator arm (138 mmol/L)
  Arms: Lower dialysate sodium
Drug: Higher dialysate sodium (142 mmol/L; using Renasol hemodialysis concentrate) — A higher dialysate sodium will be used in the experimental arm (142 mmol/L)
  Arms: Higher dialysate sodium

SUMMARY:
Intra-dialytic hypotensive (IDH) events can be defined as an abrupt decline in blood pressure that cause symptoms and/or require an intervention. They are common, affecting up to one third of maintenance HD sessions. Detrimental associations include: development of myocardial stunning, cerebral hypo-perfusion, vascular access thrombosis and greater mortality.

Rapid solute removal by HD generates temporary osmotic gradients between the intra-vascular and intra-cellular compartments, promoting trans-cellular fluid movement and resultant hypotension. Manipulation of osmotic gradients, e.g. using higher dialysate sodium (DNa), may ameliorate excess SBP decline during HD.

This study aims to assess the effects of higher (142 mmol/L) versus lower (138 mmol/L) dialysate sodium (DNa) use in adult chronic hemodialysis patients admitted to hospital on intra-dialytic blood pressure and biomarkers of cardiac ischemia.

The investigators will randomly assign subjects to higher versus lower DNa during their hospital stay, up to a maximum of six HD sessions.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HD (>90 days)
* Age ≥18y
* Informed consent
* First admission during study period.

Exclusion Criteria:

* Use of pressors
* Pre-dialysis serum sodium <=128mmol/L or > 145 mmol/L
* Pre-dialysis SBP >180 mmHg
* Intensive care stay earlier in admission
* Expected length of stay <24 hours (e.g. admission for HD access procedure)
* Acute coronary syndrome within seven days
* Acute stroke
* Institutionalized individuals
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Finnian Mc Causland, MB, MMSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Marshall MR, Wang MY, Vandal AC, Dunlop JL. Low dialysate sodium levels for chronic haemodialysis. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD011204. doi: 10.1002/14651858.CD011204.pub3. PMID 39498822

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 patients in the lower dialysate sodium arm and 2 patients in the higher dialysate sodium arm were discharged prior to the first study session.
Period: Overall Study
Arm/Group | Lower Dialysate Sodium | Higher Dialysate Sodium
Started (Started) | 69 | 70
Completed (Completed follow up) | 69 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lower Dialysate Sodium | Higher Dialysate Sodium | Total
Number analyzed (Participants) | 69 | 70 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] — Years
  years | 61 (14) | 58 (15) | 59.5 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 34 | 60
  Male | 43 | 36 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 25 | 46
  White | 38 | 34 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 69 | 70 | 139
Diabetes [Count of Participants; unit: Participants] | 36 | 39 | 75

OUTCOME MEASURES:

1. Primary Outcome: Change in Intra-dialytic Decline in Systolic Blood Pressure
Description: Pre-dialysis SBP minus lowest intra-dialytic SBP. The data table reflect the change in systolic blood pressured (SBP) assessed at up to 6 HD sessions, where the change for each session was calculated as the pre-SBP minus the lowest SBP (during the session), and the change values from the multiple sessions were then averaged for a participant.
Time Frame: Average decline in systolic blood pressure will be measured up to a maximum of six inpatient HD sessions, occurring over a two-week time period
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Lower Dialysate Sodium | Higher Dialysate Sodium
Number analyzed (Participants) | 69 | 70
mm Hg | 26 (16) | 23 (16)

2. Secondary Outcome: Change in Pre-dialysis High-sensitivity Troponin I
Description: Cardiac injury biomarkers
Time Frame: The change in pre-dialysis high sensitivity troponin I concentrations will be measured between the first and second inpatient hemodialysis sessions, occuring over a period of three days
Population: No measured due to sample storage issues
Arm/Group | Lower Dialysate Sodium | Higher Dialysate Sodium
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From randomization to maximum of 6 inpatient study sessions (two-week period)
Arm/Group | Lower Dialysate Sodium | Higher Dialysate Sodium
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/70
Serious Adverse Events (participants affected / at risk) | 1/69 | 1/70
Other Adverse Events (participants affected / at risk) | 28/69 | 24/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower Dialysate Sodium (N=69) | Higher Dialysate Sodium (N=70)
NSTEMI non-ST segment elevation myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — NSTEMI non-ST segment elevation myocardial infarction
post-operative bleed (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Post-operative bleed
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower Dialysate Sodium (N=69) | Higher Dialysate Sodium (N=70)
Hypotension (Cardiac disorders) | 9 (9) | 6 (7)
Hypertension (>180 mmHg) (Cardiac disorders) | 3 (3) | 7 (7)
Chest pain/myocardial infarction (Cardiac disorders) | 4 (4) | 1 (1)
Cramping (Musculoskeletal and connective tissue disorders) | 7 (10) | 6 (8)
Other pain (Nervous system disorders) | 5 (8) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT02145260/Prot_SAP_000.pdf